CLINICAL TRIAL: NCT03648242
Title: Improving Pediatric Obesity Practice Using Prompts (iPOP-UP): Using Electronic Health Records to Support Decision-Making in Pediatric Obesity Care
Brief Title: Improving Pediatric Obesity Practice Using Prompts
Acronym: iPOP-UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Boston Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2000026382; 1K08HS024332-01A1 (AHRQ)
Record Dates: First submitted 2018-08-21; First posted 2018-08-27 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Pediatric Obesity
Keywords: pediatric obesity; electronic health record; clinical decision support
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interruptive Clinical Decision Support (Experimental)
  Interventions: Behavioral: Interruptive Clinical Decision Support

INTERVENTIONS:
Behavioral: Interruptive Clinical Decision Support — An interruptive, "soft-stop" alert will pop up when a pediatric primary care provider open a child's electronic health record (i.e., a new window in the forefront of the screen interrupting workflow and requiring the clinician to take an action) alerting them that the child meets criteria for obesity based on their age/sex-specific BMI percentile. The pop-up alert includes:
  * One-click addition of elevated BMI to problem list
  * Reminder to utilize Suggested PowerPlan
  * One-click access to a patient handout on evidence-based behavior change goals (screen time, sugary drinks, physical activity, sleep) and link to additional handouts and resources
  * Tables displaying trends in growth measures, blood pressure and relevant laboratory tests
  * Links to existing, evidence-based childhood obesity screening and management guidelines

SUMMARY:
This study compares the effectiveness of electronic health record (EHR)-based tools to support the management of pediatric obesity in primary care. All clinicians will receive an interruptive "pop-up" alert We will examine the impact -- the added value versus unintended consequences -- of the interruptive alert on the quality of obesity management in pediatric primary care.

DETAILED DESCRIPTION:
The primary specific aims of this study are to:

1. To assess the impact of EHR-based tools for pediatric obesity in primary care. Hypotheses: EHR-based clinical decision support tools that interrupt but support clinical workflow will (1) improve measures of pediatric obesity care quality delivered by clinicians (e.g., addition of obesity to the problem list, recommended screening for comorbidities, and follow-up/referral plans) and (2) result in a reduced rate of BMI increase over one year among children with obesity.
2. To utilize a mixed methods approach with surveys and semi-structured qualitative interviews with clinicians to (1) examine the extent to which the EHR tools positively impact clinicians' awareness, knowledge and adherence to expert guidelines for pediatric obesity management, and (2) to explore the barriers to and facilitators of clinicians' use of the EHR tools and factors that influence adoption.

ELIGIBILITY:
All pediatric primary care providers providing well child care for patients ages 2-17 years-old in the Boston Children's Hospital primary care practices will be eligible for the study. There are no exclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in body mass index (BMI) | 1 year pre-intervention, baseline, and 1 year post-intervention
  change in BMI, calculated from height and weight measured as part of routine clinical practice during primary care clinic visits and documented in the EHR
Change in percent BMI above the 95th percentile (%BMIp95) | 1 year pre-intervention, baseline, and 1 year post-intervention
  Change in percentage of age/sex-adjusted BMI above the 95th percentile (%BMIp95), calculated from height and weight measured as part of routine clinical practice during primary care clinic visits and documented in the EHR
Change in documentation of elevated BMI diagnosis | 1-year pre-implementation compared to 1-year post-implementation
  Change in proportion of patients with obesity who have elevated BMI documented in the EHR
Change in proportion of patients with obesity | 1-year pre-implementation compared to 1-year post-implementation
  Change in proportion of patients with obesity who receive age-appropriate screening for comorbidities (blood measure measurement and age-appropriate laboratory screening)
Change in proportion of patients with obesity who have counseling for obesity-related behavior change documented in the EHR | 1-year pre-implementation compared to 1-year post-implementation
Change in proportion of patients with obesity with follow-up or referral orders | 1-year pre-implementation compared to 1-year post-implementation

SECONDARY OUTCOMES:
Change in provider knowledge, attitudes and practice around obesity management in primary care assessed via an electronic surveys and qualitative interviews of clinicians | baseline compared to 6 months post-implementation
System usability scale (SUS) score | 6 months post-implementation
  the system usability scale is a validated 10-item measure of system usability

CONTACTS AND LOCATIONS:
Overall Officials: Corinna Rea, MD, MPH, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No